CLINICAL TRIAL: NCT01896206
Title: CNAP Accuracy in the Bariatric Surgery Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chairman - Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB12-00808
Record Dates: First submitted 2013-06-27; First posted 2013-07-11 (Estimated); Results first posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CNAP monitor (Experimental): Subjects undergoing bariatric surgery and monitored using the CNAP monitor.
  Interventions: Device: CNAP monitor

INTERVENTIONS:
Device: CNAP monitor — Patients undergoing bariatric surgery and being monitored using the CNAP monitor.

SUMMARY:
This study will compare accuracy of a newly developed monitor for continuous non-invasive blood pressure monitoring (CNAP™ Monitor 500; CNSystems Medizintechnik AG, Graz, Austria) that provides beat-to-beat BP readings with two of the current and more commonly used intermittently oscillometric non-invasive blood pressure device (NIBP), and the invasive arterial line (IBP).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for laparoscopic bariatric surgery for the treatment of obesity
* Patients in whom an indwelling arterial cannula will be placed for the surgical procedure

Exclusion Criteria:

* Patients with history of a peripheral neurologic or neuropathic disorder
* Patients in whom an invasive arterial cannula cannot be placed
* Patients with vascular implants at the sites of non-invasive blood pressure measurement (fingers and upper arm of the examined arm)
* Edematous patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Tobias, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CNAP Monitor
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CNAP Monitor
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.55 (2.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: The Absolute Difference in Mean Arterial Pressure Between the Arterial Catheter and the CNAP.
Description: To avoid biasing the data, the absolute, not directional, difference was used. For example, if the reading from the CNAP device was 10 mmHg above or below the reading from the AC, a value of 10 mmHg was used, not -10 or +10 mmHg.
Time Frame: Participants will be followed for the duration of surgery, an expected average of 2 hours.
Population: The initial study cohort included 21 patients; however, the finger cuff was expired in 1 patient, resulting in no data collection, and the data from 2 other patients were lost in the download to the electronic medical record system.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CNAP Monitor
Number analyzed (Participants) | 18
mmHg | 7.7 (4.9)

ADVERSE EVENTS:
Arm/Group | CNAP Monitor
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes